CLINICAL TRIAL: NCT07364383
Title: Microbiome and Wellbeing Modulation in Women: An Exploratory Probiotic Study
Brief Title: Probiotics for Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cultech Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: MMS
Record Dates: First submitted 2026-01-06; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Probiotic; Microbiome; Wellbeing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): Lab4 Multi-strain Probiotic + Lactobacillus gasseri and Lactobacillus crispatus (comprising Lactobacilli and bifidobacteria species) with Vitamin A and Vitamin D
  Interventions: Dietary Supplement: Lab4 + Lactobacillus gasseri and Lactobacillus crispatus
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Lab4 + Lactobacillus gasseri and Lactobacillus crispatus — Lactobacillus acidophilus CUL-60, Lactobacillus acidophilus CUL-21, Lactobacillus gasseri CUL-09, Lactobacillus crispatus LCR15, Bifidobacterium bifidum CUL-20 and Bifidobacterium animalis subsp. lactis CUL-34 at a dose of 20 billion bacteria per/ day combined with vitamin A (800 IU/day) and Vitamin D (1000 IU/day) on a microcrystaline cellulose (MCC) base Daily dose: 20 billion bacteria per day
  Arms: Active
Other: Placebo — MCC alone
  Arms: Placebo

SUMMARY:
Investigation into the effect of probiotic supplementation on the wellbeing of women with a history of vaginal discomfort and/or irritation, along with any microbiome changes.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy menstruating women (female at birth), 18 to 40 years old with history of 3 or 4 episodes of vaginal discomfort (1 or more days) involving itching, burning sensation and/or odorous discharge in the past 12 months
2. Willing to start on completion of monthly cycle (< 5 days post completion)
3. Willing to provide vaginal and faecal samples
4. Willing to maintain normal diet and lifestyle during the study
5. Willing to refrain from taking other probiotic supplements during the study
6. Willing to refrain from sexual activity, the use of lubricants and vaginal cleaning (with antibacterials)/douching for 2 days prior to providing vaginal swabs

Exclusion Criteria:

1. Consumption of oral antibiotics within the last 2 months
2. Given birth in the last 3 months, currently pregnant or planning pregnancy
3. Currently experiencing (symptoms of) a vaginal or urinary infection
4. Immunodeficient or undergoing immunosuppressive therapy
5. Diagnosed with diabetes/cardiovascular disease/cancer/dementia

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 40 (Estimated)
Dates: Start 2026-01-09 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Changes in wellbeing through the use of wellbeing diaries | From date of randomization until the end of the intervention period (20 days)
  Changes in wellbeing and in the composition of the microbiome
Changes in microbiome composition through shotgun Metagenomics | From date of randomization until the end of the intervention period (20 days)

CONTACTS AND LOCATIONS:
Locations (1):
- Comac Medical, Sofia,, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: Yes